CLINICAL TRIAL: NCT07039253
Title: Engaging Together for Healthy Relationships Version 2.0: Multisite Pilot Intervention Trial
Brief Title: Pilot Trial of Clinic-based Dating Violence Prevention Program for Adolescents and Caregivers
Acronym: ETHR2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maya Ragavan, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY25030017; 1R21HD109627-01A1 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-05

CONDITIONS: Dating Violence; Parent; Primary Care
Keywords: dating violence prevention; parental monitoring and communication; pilot trial; middle school
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engaging Together for Healthy Relationships (Experimental): Providers and families in the intervention arm will receive the ETHR program which includes a clinician training, provider scripts, resource guides, a take home box for families, post-visit text messages, a comprehensive website, and warm referral processes.
  Interventions: Behavioral: Engaging Together for Health Relationships

INTERVENTIONS:
Behavioral: Engaging Together for Health Relationships — Dating violence intervention for caregivers and adolescents to be delivered within pediatric primary care

SUMMARY:
ETHR V 2.0 pilot trial is a one-arm, multi-site pilot trial to assess the acceptability and feasibility of Engaging Together for Healthy Relationships, a caregiver-adolescent dating violence prevention program delivered within pediatric primary care.

DETAILED DESCRIPTION:
ETHR V 2.0 pilot trial is a one-arm (intervention only) pilot trial of Engaging Together for Healthy Relationships, a caregiver-adolescent dating violence prevention program delivered within pediatric primary care. We completed one round of the pilot trial in two clinics in Pittsburgh and now are expanding the trial to include two sites with all providers in each site. ETHR includes clinician training, in-clinic resources, and after visit text messages and resources for families. This is an intervention only trial to assess acceptability, feasibility, and exploratory pre/post changes in outcomes.

ELIGIBILITY:
Inclusion Criteria

Providers:

1. Sees patient at an eligible primary care clinic
2. Speaks and understands English
3. Age 18 or older
4. Identifies as a pediatrician, nurse practitioner, physician assistant (pediatric primary care healthcare provider)

Adolescents

1. Age 12 to 16
2. Attending an upcoming well-child visit from a provider enrolled in the study
3. Caregiver who is accompanying well-child visit with adolescent is also participating
4. Speaks and understands English

Parents

1. Is parent or primary caregiver for an adolescent age 12 to 16
2. Adolescent has an upcoming well-child visit with a provider enrolled in the study
3. Accompanying child to the well-visit
4. Adolescent is interested and eligible to participate in study
5. Speaks and understand English

Exclusion Criteria:

* Unable to assent/consent
* Does not meet inclusion criteria

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who are eligible out of the total who are approached | Through completion of study recruitment, an average of 6 months
  Will assess through tracking data
Percentage of participants who are consented out of the total who are eligible | Through completion of study recruitment, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the baseline survey out of the total who consented | Through completion of completing baseline surveys, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the well-visit out of the total who consented | Through completion of completing well-visits, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the immediate post-intervention survey out of the total who consented | Through completion of completing post-intervention survey, an average of 7 months
  Will assess through tracking data
Percentage of participants who complete the 1-month post-intervention survey out of the total who consented | 4 months
  Through completion of completing 1- month post-intervention survey, an average of 8 months
Percentage of participants who complete the 3-month post-intervention survey out of the total who consented | Through completion of completing 3 month post-intervention survey, an average of 12 months
  Will assess through tracking data
Percentage of participants who strongly agree or agree that the intervention is acceptable using a 4-item validated measure (Acceptability of Intervention Measure) | Through completion of completing immediate post-visit surveys, an average of 6 months
  Validated measure (Acceptability of Intervention Measure)
Percent of participants who received intervention during pediatric primary care visit | Through completion of completing well-visits, an average of 6 months
  Investigator-developed measure with questions about what components of the intervention were received during the well visit
Participants use intervention resources after the visit | Through completion of intervention, on average 3 months post well visit
  Investigator-developed measure on use of intervention resources after the visit

SECONDARY OUTCOMES:
Self-efficacy in preventing adolescent relationship abuse (ARA), change in outcome between baseline and 3 months | Baseline, 3-month post intervention
  Self-efficacy around ARA prevention, 1-5 scale (5=higher self-efficacy)
Percentage of participants who utilize ARA resources at each measurement point, change in outcome over time | Baseline, 1 month post intervention, 3 month post-intervention
  Investigator developed measure (yes/no)
Attitudes about ARA, change in outcome between baseline and 3 months | Baseline, 3-month post intervention
  Attitudes about Abusive Relationships, 1-5 scale (1=not abusive, 5=very abusive)
Motivation around preventing dating violence | Baseline, 3-month post intervention
  Investigator developed measure, 1-5 scale (1=not motivated, 5=very motivated)
Parent-adolescent communication around dating and ARA, change in outcome over time | Baseline, 3-month post intervention
  Investigator developed measure, yes/no answer choices (yes=has communicated, no=has not communicated)
Parental monitoring around dating and ARA, change in outcome over time | Baseline, 3-month post intervention
  Investigator developed measure, 1-5 scale (1=never; 5=always)
Percentage of adolescents reporting ARA victimization and perpetration | Baseline, 3-month post intervention
  CADRI Short Form 1-5 scale (never to everyday)
ARA knowledge | baseline, 3 months surveys (6 months total)
  3 questions assessing ARA knowledge (yes/no answer choices)

CONTACTS AND LOCATIONS:
Overall Officials: Maya Ragavan, MD, MPH, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Community Practice, Monongahela, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
To protect confidentiality and due to the sensitivity of this topic, we will not share IDP